CLINICAL TRIAL: NCT01826071
Title: Comparison of Three Treatments for Lower Extremity Apophysitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Rebecca Carl, MD, Associate Professor of Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-15150
Record Dates: First submitted 2013-03-29; First posted 2013-04-08 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Osgood-Schlatter Syndrome (OSS); Sinding-Larson and Johansson Syndrome (SLJ); Sever's Disease; Apophysitis
Keywords: Osgood-Schlatter syndrome (OSS); Sinding-Larsen and Johansson syndrome (SLJ); Sever's disease; apophysitis; growth; knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Symptomatic Treatment (No Intervention): acetaminophen, NSAID, ice and relative rest
- Static Stretch (Experimental): Home exercise program with static stretching
  Interventions: Other: Static Stretch
- Active Elongation (Experimental): Home exercise program with active elongation exercises
  Interventions: Other: Active Elongation

INTERVENTIONS:
Other: Static Stretch — Standing Gastrocnemius Stretch Standing Soleus Stretch Seated Gastrocnemius Stretch Seated Soleus Stretch Hamstring Stretch Quadriceps Stretch (Standing) Quadriceps Stretch (Side Lying)
  Arms: Static Stretch
Other: Active Elongation — Mini Squat- Double Leg Mini Squat- Single Leg Prone Hip Extension with Knee Flexed 3 Position Straight Leg Raises Quadriceps Myofascial Release Heel Raises (Eccentric Strengthening) Single Leg and Double Leg Gastrocnemius Myofascial Release Calcaneal Glides
  Arms: Active Elongation

SUMMARY:
The purpose of this study is to compare three different treatments for these types of lower extremity apophysitis- Osgood-Schlatter syndrome (OSS), Sinding-Larsen and Johansson syndrome (SLJ), or Sever's disease.

The investigators hypothesize that adolescents who perform a home exercise program (HEP) consisting of active elongation exercises will have decreased pain and earlier return to sports and activities as compared to those who perform a HEP that consists of static stretching exercises or those who use symptomatic treatment with ice, acetaminophen or NSAIDs and activity modification.

DETAILED DESCRIPTION:
Osgood-Schlatter syndrome (OSS), Sinding-Larsen and Johansson syndrome (SLJ), or Sever's disease are three types of apophysitis, or secondary growth center irritation, that frequently affect children and teens. Although these conditions are common, there is very little data from high quality studies to support a particular treatment method in affected patients. The purpose of this study is to compare three different treatments for these types of apophysitis. The investigators plan to compare two types of home exercise program (HEP), one involving active elongation exercises and one utilizing static stretching, with symptomatic treatment consisting of icing, over-the-counter medications and relative rest. The investigators hypothesize that the active elongation HEP will result in improvement in pain and earlier return to athletic activities when compared to the static stretching HEP and symptomatic care. This pilot study will recruit subjects at the Ann & Robert H. Lurie Children's Hospital outpatient sports medicine and orthopaedic clinics with any of the following types of lower extremity apophysitis: OSS, SLJ or Sever's disease. Subjects will complete a baseline evaluation and questionnaire and will be randomized into one of the three treatment groups. At 2, 4, 6, and 8 weeks, subjects from all groups will use a secure website to complete an online survey to complete questions regarding current pain level, compliance with their home exercise program, if applicable, use of other forms of treatment or pain management (e.g. splinting, icing, rest from activities) and current activity level. The investigators will compare results from each group to determine which treatment(s) resulted in the largest improvements in pain scores and the highest rates of participation in sports and recreational activities.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of OSS, SLJ, or Sever's disease
* must have regular access to the Internet

Exclusion Criteria:

* history of prior treatment for OSS, SLJ, or Sever's disease
* history of previous injury to the affected joint requiring more than 1 week off of sports or activities

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2023-10 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Change in pain rating of a 5 point Likert type pain scale | 8 weeks
  The Likert-type pain scale is a self-reported pain scale asking participants to rate pain

SECONDARY OUTCOMES:
Missed time from sports/physical activities | 8 weeks
  Missed time from sports/physical activities in days

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Carl, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States